CLINICAL TRIAL: NCT03825276
Title: Metabolic Adaptations and Role of Nutritionally-Mediated Gut Microbiota Changes Following Mango Consumption in Overweight Men and Women : The MANGO Pilot Study
Brief Title: Effect of Mango on Gut Microbiota and Metabolic Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Charles Couillard, Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MANGO 2018-147
Record Dates: First submitted 2019-01-22; First posted 2019-01-31 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Gut Microbiota; Metabolic Syndrome
Keywords: Mango; Polyphenols; Inflammation; Insulin resistance; Transcriptomic; Metabolomic; Metagenomic
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mango consumption (Experimental)
  Interventions: Dietary Supplement: Mango consumption

INTERVENTIONS:
Dietary Supplement: Mango consumption — Daily consumption of 280 g of frozen mangos during 8 weeks. The daily dose in equivalent to a 2-cups serving.

SUMMARY:
Mango is rich in bioactive compounds such as dietary polyphenols and carotenoids, which may explain its beneficial effect on health. Polyphenols accumulate in the gut where they can positively modulate the microbiota. As gut microbiota may have a strong influence on cardiometabolic health, we hypothesize that mango consumption improves metabolic profile in overweight or obese individuals through beneficial changes in gut microbiota. The study of metagenomics, transcriptomics and metabolomics will be used to validate this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and premenopausal women
* At least one of the following : BMI between 25 and 40 kg/m2 or Waist circumference ≥ 80 cm for women and ≥ 94 cm for men
* At least one of the following : TG ≥ 1.35 mmol/L or fasting insulinemia ≥ 42 pmol/L
* Caucasian origin

Exclusion Criteria:

* Nicotine use
* Metabolic disorders or use of medication that may affect parameters measured in the study
* Use of dietary supplements or natural health product that may affect parameters measured in the study
* Use of antibiotics in the last 3 months
* Surgery in the last 3 months or planned during the study timeline
* Alcohol consumption >2 drinks/day
* Weight change >5% in the last 3 months
* Mango aversion, allergy or intolerance
* Dietary restrictions (vegetarian, gluten avoidance...)
* Berries consumption >1 serving/day
* Pregnancy, breastfeeding or pregnancy planned within 3-6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma insulin concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma glucose concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma triglycerides concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma total cholesterol concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma HDL cholesterol concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma LDL cholesterol concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks

SECONDARY OUTCOMES:
Changes in waist circumference of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in hip circumference of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in waist to hip circumference ratio of overweight/obese men and women taking frozen mangos daily | 8 weeks
  Waist and hip circumference will be combined to report waist to hip ratio
Height of overweight/obese men and women taking frozen mangos daily | Baseline
Changes in weight of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in body mass index (BMI) of overweight/obese men and women taking frozen mangos daily | 8 weeks
  Weight and height will be combined to report BMI
Changes in systolic blood pressure of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in diastolic blood pressure of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in insulin secretion of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in insulin sensitivity of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in glycated hemoglobin (HbA1c) in overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma tumor necrosis factor (TNF-alpha) concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma interleukin-6 (IL-6) concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma high-sensitivity C-reactive protein (hs-CRP) concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in gene expression in peripheral blood mononuclear cells (PBMC) of overweight/obese men and women taking frozen mangos daily | 8 weeks
  Gene-level expression from >20,000 annotated genes will be examined
Changes in plasma metabolites concentration in overweight/obese men and women taking frozen mangos daily | 8 weeks
  Metabolites include acylcarnitines, glycerophospholipids, sphingolipids, sugars, amino acids, biogenic amines
Changes in gut microbiota composition in overweight/obese men and women taking frozen mangos daily | 8 weeks
  Stool samples will be collected and whole metagenome shotgun sequencing analysis will be conducted
Changes in plasma lipopolysaccharide (LPS) concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks
Changes in plasma LPS binding protein (LBP) concentration of overweight/obese men and women taking frozen mangos daily | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles.Couillard@fsaa.ulaval.ca Couillard, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada

REFERENCES:
- [Derived] Keathley J, de Toro-Martin J, Kearney M, Garneau V, Pilon G, Couture P, Marette A, Vohl MC, Couillard C. Gene expression signatures and cardiometabolic outcomes following 8-week mango consumption in individuals with overweight/obesity. Front Nutr. 2022 Aug 11;9:918844. doi: 10.3389/fnut.2022.918844. eCollection 2022. PMID 36034894
- [Derived] Keathley J, Kearney M, Garneau V, Toro-Martin J, Varin TV, Pilon G, Couture P, Marette A, Vohl MC, Couillard C. Changes in systolic blood pressure, postprandial glucose, and gut microbial composition following mango consumption in individuals with overweight and obesity. Appl Physiol Nutr Metab. 2022 May;47(5):565-574. doi: 10.1139/apnm-2021-0637. Epub 2022 May 4. PMID 35506190